CLINICAL TRIAL: NCT05600114
Title: A Randomized, Double-Blind, Parallel Group, Placebo-Controlled Study, Evaluating the Efficacy, Safety, and Tolerability of Cannabidiol Oral Solution in Subjects With Social Anxiety Disorder
Brief Title: Cannabidiol (CBD) for the Treatment of Social Anxiety Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: EmpowerPharm Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EPI-CBD-001
Record Dates: First submitted 2022-10-26; First posted 2022-10-31 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Social Anxiety Disorder
MeSH Terms: conditions — Phobia, Social | interventions — Cannabidiol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cannabidiol (CBD) Oral Solution 300 mg/day (Experimental)
  Interventions: Drug: Cannabidiol oral solution
- Cannabidiol (CBD) Oral Solution 600 mg/day (Experimental)
  Interventions: Drug: Cannabidiol oral solution
- Placebo Oral Solution (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cannabidiol oral solution — CBD 150 mg BID
  Arms: Cannabidiol (CBD) Oral Solution 300 mg/day
Drug: Cannabidiol oral solution — CBD 300 mg BID
  Arms: Cannabidiol (CBD) Oral Solution 600 mg/day
Drug: Placebo — Placebo BID
  Arms: Placebo Oral Solution

SUMMARY:
A phase 2, multicenter, double-blind, parallel group, placebo-controlled, randomized clinical study, designed to compare the efficacy, safety, and tolerability of 2 dose levels of CBD and a matching placebo for the treatment of subjects with Social Anxiety Disorder (SAD).

ELIGIBILITY:
Inclusion Criteria:

* Clinically predominant diagnosis of Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) SAD
* LSAS score of 70 or higher
* Females of childbearing potential must test negative for pregnancy and agree to use a reliable birth control method. Male subjects must also agree to use highly effective methods of contraception.
* Read, understand, and sign the informed consent form.
* No significant physical health abnormalities based on physical exam, ECG and laboratory tests.

Exclusion Criteria:

* Other current psychiatric disorder as the clinically predominant diagnosis.
* Lifetime diagnosis of schizophrenia or any other psychosis, MDD with psychotic features, intellectual disability, autism spectrum disorders, bipolar disorder type 1, and cannabis use disorder
* Previous 6 months diagnosis of Post-traumatic stress disorder, obsessive compulsive disorder, moderate to severe alcohol use disorder, and substance abuse disorder (except tobacco use disorder or mild alcohol use disorder)
* Severe MDD
* Use of oral psychoactive medications or beta adrenergic antagonists in the past 4 weeks, or depot neuroleptics within 12 weeks
* Electroconvulsive therapy within 6 months, psychotherapy or transcranial magnetic stimulation within 3 months
* Clinically significant abnormality or clinically significant unstable medical condition
* Impaired liver function
* Significant risk of suicide or homicide
* Pregnancy/lactation
* Sensitivity to CBD or excipients
* Current cannabis use; past frequent cannabis use
* Illegal drug use

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 239 (Actual)
Dates: Start 2022-10-27 (Actual); Primary Completion 2023-12-13 (Actual); Study Completion 2023-12-13 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline to endpoint in the Liebowitz Social Anxiety Scale (LSAS) | 10 weeks

CONTACTS AND LOCATIONS:
Locations (17):
- United States (17):
  - EPI-CBD-001 Site, Encino, California
  - EPI-CBD-001 Site, Lemon Grove, California
  - EPI-CBD-001 Site, Los Alamitos, California
  - EPI-CBD-001-Site, Oceanside, California
  - EPI-CBD-001 site, San Jose, California
  - EPI-CBD-001 Site, Jacksonville, Florida
  - EPI-CBD-001 Site, Lauderhill, Florida
  - EPI-CBD-001 Site, Maitland, Florida
  - EPI-CBD-001 Site, Orlando, Florida
  - EPI-CBD-001 Site, Chicago, Illinois
  - EPI-CBD-001 Site, Cedarhurst, New York
  - EPI-CBD-001-Site, New York, New York
  - EPI-CBD-001-Site, Rochester, New York
  - EPI-CBD-001 Site, Oklahoma City, Oklahoma
  - EPI-CBD-001 Site, Portland, Oregon
  - EPI-CBD-001 site, Wichita Falls, Texas
  - EPI-CBD-001 Site, Bellevue, Washington